CLINICAL TRIAL: NCT07015723
Title: The Correlation Between MRCP and Biopsy Pre-LDLT for Liver Steatosis Assessment: an Ambidirectional Cohort Study
Brief Title: Steatosis Assessment Pre-LDLT
Acronym: SILDLT
Status: Enrolling by invitation | Type: Observational
Sponsor: Erasmus Medical Center (Other)
Responsible Party: Principal Investigator, Robert Minnee, Hepato-Pancreato-Biliary/Transplant Surgeon, PhD, Erasmus Medical Center
Other Study IDs: 14060
Record Dates: First submitted 2025-06-04; First posted 2025-06-11 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-06

CONDITIONS: Living Donor Liver Transplantation
Keywords: Liver Transplantation; Living Donor; Magnetic Resonance Imaging; Biopsy; Anatomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Living liver donors: The population consists of adult living liver donors at the Erasmus MC.
  Interventions: Procedure: Living liver donors

INTERVENTIONS:
Procedure: Living liver donors — Adults who are screened for living liver donation.

SUMMARY:
There is a major shortage of donor livers in the Netherlands. Living donor liver transplantation (LDLT) is a good solution to this shortage. Donor screening is extensive to minimalize risks for donors and recipients. During screening, the vascular anatomy of the liver is assessed with CT, the bile duct anatomy with MRCP, and liver steatosis with a biopsy. Biopsy is an invasive intervention with some risk of complications. MRCP can aid in steatosis assessment. Previous research suggested that biopsy can be performed on indication. However, the sensitivity of detecting different steatosis percentages on MRCP varies widely, which makes determining the degree of steatosis difficult and less reliable. This project investigates whether MRCP is equally adequate as biopsy in assessing liver steatosis. It may lead to a faster, less burdensome and minimal invasive screening process.

DETAILED DESCRIPTION:
Research methods:

General and biopsy data (liver steatosis percentage) and MRCP images will be extracted from HiX. Screenshots of the images will be made. All personal data will be blacked out using Microsoft Powerpoint 16.90.2. The MRCP-images and biopsy data will be coded at random with different codes for the MRCP and biopsy of the same donor. The coded images will be shared with the radiologist through Castor. He will assess liver steatosis on MRCP. He will register his findings in Castor and share this file with the study coordinator.

Analysis:

Normality will be tested using the Shapiro-Wilk test. Homogeneity of variances will be tested using the F-test. A QQ-plot will be used to check for outliers. For the baseline donor characteristics, sex differences will be investigated for age, weight, height, and BMI using the unpaired samples t-test or Mann-Whitney test.

Similarities and differences between liver steatosis assessment on MRCP and biopsy will be thoroughly described.

The mean (Standard Deviation (SD)) percentage of liver steatosis will be calculated for MRCP and for biopsy. The correlations between MRCP and biopsy will be calculated by the following formula: (mean percentage on MRCP)/(mean percentage on biopsy)*100(%). For the mean correlation, the average of all donors' correlations will be taken. A table showing the means (SD) and min-max of the percentage of liver steatosis, and the correlation will be made. The distribution of correlations will be shown in a bar chart. The paired samples t-test will be used to test for differences in the mean percentage of liver steatosis on MRCP and biopsy. Subgroup analyses will be carried out for sex, age, weight, height, and BMI using the unpaired samples t-test, Welch's t-test, or Mann-Whitney test Statistical analyses will be carried out using RStudio 2024.09.1, GraphPad Prism 9.5.0, and Microsoft Excel version 16.90.2. P<0.05 indicates statistical significance.

Recruitment and informed consent procedures The transplant coordinator and/or transplant surgeon will inform participants about the study and will ask their written informed consent. Living liver donors are followed up annually for life. The participants will be informed during a follow-up consult. All donors who are, for whatever reason, not visiting the Erasmus MC anymore for follow-up are contacted by phone. If the donor considers participating, a Patient Information Form (PIF) will be sent by mail. The donors can return the signed PIF through mail.

Donors can withdraw their informed consent at any time and for any reason if they wish to do so without any consequences. They can withdraw through phone, mail, or in person.

Privacy protection Subject's privacy is protected by using coded data. In the database subjects are referred to as numbers. These numbers are chosen at random. Which number belongs to which subject is registered in a key table with a password. This password is only known by the principal investigator and the research team. The database in which the data is stored (Castor), meets the requirements set for data security. The handling of personal data is in compliance with the Dutch Data Protection Act (in Dutch: 'Algemene Verordening Gegevensbescherming (AVG)). Only the code number will be used for study documentation, progress reports, and research publications.

ELIGIBILITY:
Inclusion Criteria:

* Living liver donation between May 2004 and June 2026 at the Erasmus MC
* Written informed consent

Exclusion Criteria:

- There are no exclusion criteria for this study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population consists of adult living liver donors at the Erasmus MC.
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Liver steatosis | Preoperative during screening for living liver donation.
  The primary outcome is the percentage of liver steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Robert C. Minnee, MD, PhD, Principal Investigator — Erasmus Medical Center
Locations (1):
- Erasmus Medical Center, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Study protocol, documentation, data management plan, data analysis plan, script to assess data, scripts to analyse data, scripts to generate tables and figures in the publication.
Supporting Information: Study Protocol, SAP, CSR, Analytic Code
Time Frame: (Underlying) data will be made available alongside with the publication. It will be available for 10 years. Access to the data and images is approved by the head of department and principal investigator. This access is temporarily. To whom and when access approved is registered.
Access Criteria: The PI will verify the authenticity of the requesting researcher and will check whether their intentions are in line with the informed consent and whether the intended methodology is suitable and will approve the request before providing access to the data. Other researchers could express their interest in the dataset through countersigned DTA. After meeting the sharing and reuse conditions as described above and approval of the PI, data access will be provided through the data repository.

REFERENCES:
- [Background] Testa G, Nadalin S, Klair T, Florman S, Balci D, Frola C, Spiro M, Raptis DA, Selzner M; ERAS4OLT.org working group. Optimal surgical workup to ensure safe recovery of the donor after living liver donation - A systematic review of the literature and expert panel recommendations. Clin Transplant. 2022 Oct;36(10):e14641. doi: 10.1111/ctr.14641. PMID 35258132
- [Background] Yim SH, Kim DG, Kang M, Koh HH, Choi MC, Min EK, Lee JG, Kim MS, Joo DJ. Survival benefit of living-donor liver transplantation in patients with a model for end-stage liver disease over 30 in a region with severe organ shortage: a retrospective cohort study. Int J Surg. 2023 Nov 1;109(11):3459-3466. doi: 10.1097/JS9.0000000000000634. PMID 37565633
- [Background] Jackson WE, Malamon JS, Kaplan B, Saben JL, Schold JD, Pomposelli JJ, Pomfret EA. Survival Benefit of Living-Donor Liver Transplant. JAMA Surg. 2022 Oct 1;157(10):926-932. doi: 10.1001/jamasurg.2022.3327. PMID 35921119
- [Background] Ter Burg HW, Chorley Rn AJ, Polak WG, Kranenburg LW, Boehnert MU, Minnee RC. Older living liver donors can enlarge the donor pool: a systematic review and meta-analysis. Int J Surg. 2024 Aug 1;110(8):5022-5033. doi: 10.1097/JS9.0000000000001419. PMID 38573086